CLINICAL TRIAL: NCT05371704
Title: The Effect of Micronutrient Supplementation on Gut Microbiome Composition and Function
Acronym: Multigut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Professor, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Version 1
Record Dates: First submitted 2022-02-03; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Gastrointestinal Microbiome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation (Experimental): In this arm of the study, participants will take 1 multivitamin pill each day for 10 days. If this is the participant's first trial, they will also record their diet in a 10-day estimated food diary. If this is the participant's second trial, they will replicate their diet recorded from their first trial.
  Interventions: Dietary Supplement: Multivitamin Supplementation; Other: Dietary Replication
- Control (Other): In this arm of the study, participants will not supplement with any multivitamin. If this is the participant's first trial, they will record their diet in a 10-day estimated food diary. If this is the participant's second trial, they will replicate the diet recorded from their first trial.
  Interventions: Other: Dietary Replication

INTERVENTIONS:
Dietary Supplement: Multivitamin Supplementation — Participants will supplement daily with an over-the-counter oral multivitamin pill
  Arms: Supplementation
Other: Dietary Replication — Patients will record their dietary intake in an estimated food diary during the first trial. During the second trial, participants will be asked to replicate their diet from the first trial

SUMMARY:
The main aim of this randomized crossover study is to explore the effect of micronutrient supplementation on gut microbiota composition and function in healthy volunteers. Participants will undertake two 10-day trials with a replicated diet separated by a 15-day washout period. For one of these trials, participants will take a daily over-the-counter multivitamin supplement. Faecal and urine samples will be collected at the start and end of each trial to assess changes in gut microbiota composition, urinary and faecal metabolomics, and targeted bacterial metabolites including short chain fatty acids, sulphide, and lactate.

DETAILED DESCRIPTION:
Exploring the effect of habitual dietary patterns on human gut microbiota and on host health is an area of scientific interest and a major funding theme in UKRI. The main aim of this proof-of-concept study is to explore the effect of micronutrient supplementation on gut microbiota composition and function in healthy volunteers.

Participants will be asked to undertake two trials with 15 day washout in-between. If the participants are allocated to the "supplementation group" they will be asked to consume an over-the-counter multivitamin supplement for 10 days (1 tablet per day) in addition to their usual diet. Participants will provide faecal and urinary samples prior to initiation of the intervention and again at the end of the 10-day supplementation. During these 10 days participants will be asked to record the meals they consume on provided food diaries. If the participants are allocated to the "control group", participants will be asked to provide the same number of samples and at the same intervals as the supplementation group (i.e. at baseline and after 10 days) but without receiving micronutrient supplementation. Participants will also be asked to replicate as close as possible the diet they had followed during the first trial they were allocated. Between the two trials, participants will follow a wash-out period of 15 days with the aim of reverting the gut microbiota characteristics back to baseline levels.

The main outcome measures of this study are to assess changes in gut microbiota composition based on 16S rRNA gene amplicon sequencing, changes in urinary/faecal metabolomics, and changes in targeted bacterial metabolites (short chain fatty acids, sulphide, lactate).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults >18 y

Exclusion Criteria:

* History of previous major gut surgery,
* Unstable weight,
* Use of pre/probiotics, micronutrient supplements, antibiotics, or steroids the last 3 months
* Participation in other research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota composition during multivitamin supplementation | This will be assessed 4 times throughout the study. This will be assessed at the beginning (day 0) and end (day 10) of each 10-day trial.
  Changes will be assessed via 16S rRNA gene amplicon sequencing from DNA extracts of faecal samples
Changes in concentrations of faecal and urinary metabolites during multivitamin supplementation | This will be assessed 4 times throughout the study. This will be assessed at the beginning (day 0) and end (day 10) of each 10-day trial.
  Concentration of several urinary and faecal metabolites will be assessed via 1H NMR spectroscopy in urine and faecal samples from study participants. Changes during multivitamin supplementation will be investigated.
Changes in bacterial metabolites during multivitamin supplementation | This will be assessed 4 times throughout the study. This will be assessed at the beginning (day 0) and end (day 10) of each 10-day trial.
  Changes in targeted bacterial metabolites including short chain fatty acids, sulphide, ammonia, lactate, succinate, ethanol

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, University of Glasgow / New Lister Building, Glasgow Royal Infirmary, Glasgow, United Kingdom

REFERENCES:
- [Derived] Mckirdy S, Koutsos A, Nichols B, Anderson M, Dhami S, Chowdhury CR, Mascellani Bergo A, Havlik J, Gerasimidis K. Micronutrient supplementation influences the composition and diet-originating function of the gut microbiome in healthy adults. Clin Nutr. 2025 Aug;51:293-303. doi: 10.1016/j.clnu.2025.06.020. Epub 2025 Jun 25. PMID 40645132